CLINICAL TRIAL: NCT04873401
Title: Leveraging Social Networks to Increase COVID-19 Testing Uptake: A Comparison of Credible Messenger and Chain Referral Recruitment Approaches
Brief Title: Leveraging Social Networks to Increase COVID-19 Testing Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Alliance for Postive Change (Other); Argus Community Inc. (Other); Columbia University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Katherine Elkington, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 8153; UG1DA050071-04S1 (NIH)
Record Dates: First submitted 2021-03-24; First posted 2021-05-05 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Covid-19; Substance Use; Opioid Use
MeSH Terms: conditions — COVID-19; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Groups are randomly assigned to either condition/arm; after 6 months they each cross over into the other arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chain Referral (Experimental): In the chain-referral intervention, a discrete number of "seeds" will be recruited from the community partners, trained and incentivized to recruit and refer members of their social networks to receive COVID-19 testing; these recruits are then trained to do the same.
  Interventions: Behavioral: Chain-referral
- Credible Messenger (Experimental): In the credible messenger intervention, peers identified as popular and socially influential individuals within their respective communities with lived experience are trained to engage within formal and informal social networks to promote behavior change.
  Interventions: Behavioral: Credible Messenger

INTERVENTIONS:
Behavioral: Chain-referral — In the chain-referral intervention, a discrete number of "seeds" will be recruited from the community partners, trained and incentivized to recruit and refer members of their social networks to receive COVID-19 testing. The peer recruiters are paid for each suvcessful and eligible recruit who enrolls to be tested. Those individuals are then themselves trained to recruit peers from their social networks to receive COVID-19 testing. This is repeated over a period of 4-6 months.
  Arms: Chain Referral
Behavioral: Credible Messenger — In the credible messenger intervention, peers noted to be popular and socially influential individuals with lived experience will be trained to engage within community settings and areas to encourage community members to receive COVID-19 testing at the community partnering agencies. Peers will recruit community members over a period of 4-6 months.
  Arms: Credible Messenger

SUMMARY:
This two-year project will adapt and conduct a trial examining the ability of two recruitment strategies, chain-referral and credible messenger, to reach those who use opioids and other substances in order to increase their uptake of onsite point of care COVID-19 testing that will be delivered in two community based organizations (CBOs): Alliance for Positive Change and Argus Health Inc. In Phase 1, Adapt two implementation strategies to support COVID-19 testing uptake and sustainability, adapting elements of existing efficacious social network-based interventions via a CBPR approach. In Phase 2, we will examine and compare the efficacy of two sets of implementation strategies on (i) reach, (ii) testing uptake, (iii) service delivery (i.e. quarantine, medical care, contact tracing) and (iv) sustainability for individuals who use opioids and other drugs. In Phase 3, Elucidate and compare the system/organizational-, staff-, and individual-level factors that influence implementation (i.e. fidelity, acceptability, feasibility, sustainability) of the strategies to develop a plan for dissemination and scale-up in other CBOs who serve opioid and other substance using individuals in NYC.

DETAILED DESCRIPTION:
Aims. Building on the expertise and community out-reach infrastructure of two community-based organizations (CBOs), Argus Community Inc. and Alliance for Positive Change, and following a CBPR approach, investigators propose to take two implementation strategies that have been proven to increase the reach, access, and uptake of HIV testing and related services, and adapt them to support the uptake and sustainability of point-of-service (POS) onsite COVID-19 testing in CBOs that target the underserved population of those who use opioids and other substances. Guided by social cognitive theory, Andersen's model of health care access and the EPIS framework, the specific aims are to:

(1). Adapt two implementation strategies to support COVID-19 testing uptake and sustainability, adapting elements of existing efficacious social network-based interventions via a CBPR approach; (2). Examine and compare the efficacy of two sets of implementation strategies on (i) reach, (ii) testing uptake, (iii) service delivery and (iv) sustainability for individuals who use opioids and other drugs. Use of data drawn from Healthix, a public health information exchange, will supplement this comparison by generating a baseline of participant prior testing and health behavior to determine access to underserved populations as well as long-term influence on future testing behavior; and (3) Elucidate and compare the system/organizational-, staff-, and individual-level factors that influence implementation of the strategies to develop a plan for dissemination and scale-up in other CBOs who serve opioid and other substance using individuals in NYC.

Settings. Alliance for Positive Change and Argus Health Inc have well-established partnership with members of the parent grant team following partnerships on numerous initiatives targeting HIV, HCV and STIs prevention, testing and treatment for over 20 years. Argus and Alliance have had a combined presence in the communities of Washington Heights, Harlem and the South Bronx for over 50 years, and have subsequently developed considerable trust, support and "credibility" within these communities.

Design, Sample Size and Randomization. Two distinct social network recruitment strategies will be adapted and compared. Guided by the EPIS framework, SCT, and Andersen's Model, this 2-year study will comprise three phases. In Phase 1: Adaptation of outreach recruitment strategies, investigators will work with our project CAB, via a CBPR approach, to adapt chain-referral and POL strategies for uptake of COVID-19 testing, to finalize recruitment and on-site testing protocols. In Phase 2: Strategy Efficacy Trial and Implementation Evaluation, investigators will compare the two strategies in a cross-over design at two CBOs, with initial strategy assignment randomly determined and rolled out for 4 months before cross-over. Investigators will examine the impact of each strategy on (i) reach, (ii) COVID-19 testing/repeat testing, and (iii) service delivery among those who test positive for COVID-19. In Phase 3: Sustainment, CBOs will implement the strategy with more favorable outcomes in Phase 2, and investigators will examine their sustainment of the program. Implementation evaluation will identify participant-, staff-, and organizational-level factors that influence the feasibility, acceptability, and sustainability of each strategy in the CBOs.

Phase 1: Adaptation of Outreach Strategies. Investigators will employ a CBPR-guided approach to adapt the social network-based outreach strategies. To do this, investigators will hold four 1-hour working groups with our CAB. All CAB members will be reimbursed for their time. These groups will address how to best employ the different strategies to reach our target population and motivate testing uptake. Protocols will be shaped by findings from working group meetings and shared back to the CAB who will provide feedback to inform changes in content and format, and help identify markers of success and potential challenges.

Phase 2: Strategy Efficacy Trial and Implementation Evaluation Overview. During the first 4 months of Phase II each site will roll out a different recruitment strategy (randomly assigned 1:1) to the site Following four months of implementation, the sites will conduct a rapid PDSA through a series of four, weekly workgroups. Revisions to protocols will be made during these meetings and then the sites will "cross-over" and implement the other recruitment strategy for the next four months. Participants may be recruited twice, once in each strategy; any instances of repeat testing will be documented.

Participants. In Phase 2, using two different strategies, investigators aim to enroll N=500 individuals with a history of opioid and/or substance abuse within the past 6 months. Based on the geographic catchment areas of Argus and Alliance and current demographics of their current substance using clientele, investigators anticipate participants will be 64% male, 51% African American, 39% Hispanic. Inclusion/exclusion criteria. All participants, regardless of recruitment strategy, must endorse opioid or other substance abuse in the past 6 months, and must speak English or Spanish; >18years.

Study enrollment, and consent. Once an individual is screened at the agency and determined to be eligible, Research Assistants (RAs) will obtain written informed consent for study participation and consent to access their clinical information in Healthix, a large health information exchange in NYC. Following consent, the RA will administer the baseline assessment in a private office. Participants will receive remuneration in accordance with standards in this population. These procedures will occur in the same way regardless of recruitment method into the study.

Strategy Efficacy Trial and Implementation Evaluation. Chain-referral Strategy. Recruitment of seed participants. N=16 participants who meet inclusion criteria will be recruited from among clients at Argus and Alliance (n=8 at each site) to serve as seeds. Seeds will be stratified by substance use treatment status and gender. Site staff will contact selected individuals and refer those interested to the research team who will screen for eligibility. Following the completion of the screen, the participant will be offered COVID-19 testing; they will be compensated $20 for completing the interview at the end of the visit. Participants will be given the option to help recruit others to receive a COVID-19 test for a small incentive. If participants agree, they will receive a brief training on recruitment and three coupons. The participants will be instructed to give these coupons only to people they know who use substances.

Chain-referral recruitment: Individuals redeeming coupons will be screened for study participation, assessed and offered COVID-19 testing. Those eligible and interested will be enrolled. Procedures for informed consent, study enrollment and peer education training will be identical to those for seeds. Participants will return after three weeks to receive a recruitment incentive of $10 for every coupon redeemed. During this second visit they will complete a brief questionnaire to quantify peer-recruitment attempts.

Sample size: All participants will receive a maximum of four coupons to prevent the development of "professional recruiters." The process will continue until the sample size exceeds 125 persons (at each site) or the recruitment period is over. Based on prior work with similar populations in NYC investigators anticipate being able to recruit 125 participants for a COVID-19 test in 16 weeks.

POL Strategy: Alliance and Argus have existing POL/peer outreach programs with well-established histories of community involvement. Investigators will leverage this existing infrastructure and adapt to focus on COVID-19 testing. Based on protocols developed in Phase 1, POLs will be trained to (i) initiate conversations related to stopping transmission of COVID-19; (ii) deliver effective messages endorsing benefits of COVID-19 testing, social distancing and mask wearing; (iii) identify and visit those venues known to them where those with substance use will likely congregate; (iv) set goals to engage in conversations about COVID-19 testing with the target population and (v) document/track efforts.

Recruitment of participants via credible messengers: Based on these organizations' previous POL recruitment, 4 POLs are able to recruit 10 participants per week for HIV testing and related services. This will permit recruitment of 3-4 participants/week per POL (12-16 total/week), allowing completion of enrollment for outreach strategy in 4 total months. Participants recruited via POL will be consented and interviewed in the same manner as described above. Following the interview, participants will then be offered COVID-19 testing; they will be compensated $20 for completing the interview.

Quality Improvement (QI)/PDSA: Following the completion of the first 4-month recruitment period, agency staff, CAB members and POLs will participate in quality improvement. Using an abbreviated PDSA protocol, stakeholders across both agencies will participate to facilitate information sharing, cross-learning, and capacity building. They will refine messaging, procedures, and educational content, and make a plan to implement change during the next recruitment period. The fourth workgroup will address issues associated with internal site logistics.

Assessment and analysis. Investigators will examine the impact of the intervention on (i) reach, (ii) testing uptake and (iii) service delivery; and (iv) sustainability for individuals who use opioids and other drugs as well as potential mediating/moderating variables from the Andersen, SCT and EPIS models. Data drawn from Healthix on prior and future COVID-19 testing will augment study data to determine access to underserved populations and influence on future testing behavior.

Implementation assessment. A multi-method approach will allow us to identify implementation features that promote optimal testing uptake in the context of these CBOs. To quantify implementation, investigators will conduct staff survey assessments, monthly process checklists and a focus group.

Staff recruitment for surveys and focus groups. Staff will be eligible if they are currently employed at either Argus or Alliance, including POLs participating in Peer programs. Considerable effort will be taken to ensure that staff do not feel coerced to participate. Staff and organizational-level EPIS-derived factors will be assessed the launch of the testing initiative and after 12 months.

Monthly process assessments. Once the recruitment strategy protocols are finalized, investigators will develop the following monthly process assessments to be completed by agency staff and POLs. Feasibility: Investigators will develop a strategy specific feasibility checklist measuring three types of program delivery obstacles: obstacles to target population participation; concrete obstacles; and site/staffing obstacles. Fidelity: To assess the relationship between planned and actual implementation, investigators will design a checklist-based monitoring system with assessments completed by POLs and agency staff after a) testing/screening, b) education of recruits; recruits will also complete a brief checklist that documents time and effort in recruiting chains. Acceptability and Sustainability: Investigators will assess qualitatively implementation challenges to acceptability and sustainability via a series of two implementation focus groups with agency staff and POLs following completion of the project.

Analysis overview and main outcomes. The primary outcome of interest comparing the strategies will be testing occurrence as an indicator of testing uptake. An important secondary outcome will be reach measured through the number of coupons redeemed.

ELIGIBILITY:
Inclusion Criteria:

* Endorse opioid use in the past 6 months
* Speak English or Spanish
* Age 18+

Exclusion Criteria:

* Deny history of opioid use (but will be offered COVID-19 testing)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Elkington, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chain Referral | Credible Messenger
Started | 271 | 227
Completed | 263 | 223
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Population: The number of participants who were eligible and enrolled in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Chain Referral | Credible Messenger | Total
Number analyzed (Participants) | 263 | 223 | 486
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 254 | 217 | 471
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (9.5) | 46.8 (10.1) | 47.3 (9.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 191 | 166 | 357
  Gender: Female | 66 | 51 | 117
  Gender: Non-binary/other | 4 | 6 | 10
  Gender: Prefer not to answer | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latinx | 196 | 142 | 338
  White (non-Hispanic) | 25 | 33 | 58
  Black (non-Hispanic) | 34 | 38 | 72
  Other (non-Hispanic) | 7 | 5 | 12
  Unkown | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 263 | 223 | 486

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Agreed to Take a COVID-19 Rapid Test of Those Enrolled
Description: Number of participants who agreed to take a COVID-19 rapid test out of those who were enrolled (n=498)
Time Frame: Baseline
Measure: Number; unit: participants who tested
Arm/Group | Chain Referral | Credible Messenger
Number analyzed (Participants) | 271 | 227
participants who tested | 261 | 214
Statistical Analysis 1: Comparison: Chain Referral vs Credible Messenger; Test type: Superiority; p = 0.928, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.39 to 2.79], Standard Error of Mean 0.49

2. Primary Outcome: Mean Number of COVID-19 Rapid Tests Taken
Description: Mean number of COVID-19 rapid tests taken among those who took at least 1 test (n=478)
Time Frame: Baseline
Population: Among those who took any COVID-19 test
Measure: Mean (Standard Deviation); unit: mean number of tests taken
Arm/Group | Chain Referral | Credible Messenger
Number analyzed (Participants) | 261 | 217
mean number of tests taken | 1.8 (1.75) | 1.6 (1.35)
Statistical Analysis 1: Comparison: Chain Referral vs Credible Messenger; Test type: Superiority; p = 0.240, Regression, Linear; Median Difference (Final Values) = -0.173, 95% CI 2-sided [-0.24 to 0.115], Standard Error of Mean 0.147

3. Primary Outcome: Uptake of the Recruitment Strategy Into the Community
Description: Total number of coupons redeemed (Chain referral arm) out of coupons delivered OR total number of people approached in the community via credible messengers (Credible messenger arm) who enrolled in the study
Time Frame: Baseline
Population: Number of people who were recruited via either CM or CR strategy
Measure: Count of Participants; unit: Participants
Arm/Group | Chain Referral | Credible Messenger
Number analyzed (Participants) | 654 | 409
Participants | 271 | 227
Statistical Analysis 1: Comparison: Chain Referral vs Credible Messenger; Test type: Superiority; p = 0.367, Regression, Linear; Slope = 0.1171, 95% CI 2-sided [0.05 to 0.29], Standard Error of Mean 0.062

4. Primary Outcome: Reach of the Recruitment Strategy Into the Community
Description: Number of people reached or approached via coupon (CR) based on number of coupons distributed or via peer/direct contact (CM), who may or may not have enrolled in the study
Time Frame: Baseline
Population: The population is greater than those enrolled as this is the total number of people approached in the community. Not all people approached/recruited were enrolled into the study. Nonetheless, determining the difference in recruitment yield was a key part of the study goals.
Measure: Number; unit: people approached
Arm/Group | Chain Referral | Credible Messenger
Number analyzed (Participants) | 624 | 468
people approached | 624 | 468
Statistical Analysis 1: Comparison: Chain Referral vs Credible Messenger; Test type: Superiority; p = 0.005, Regression, Linear; Slope = 0.171, 95% CI 2-sided [0.05 to 0.29], Standard Error of Mean 0.062

5. Secondary Outcome: Participant Acceptability of Recruitment Strategy and Testing Program Scale
Description: Scale developed for study to assed ranked participant perceived acceptability of elements of the recruitment strategy and testing experience
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2025-10

6. Secondary Outcome: Sustainability of the Testing Program
Description: Number of tests conducted after the Implementation phase
Time Frame: Sustainment
Reporting Status: Not Posted

7. Secondary Outcome: Feasibility of Recruitment and Testing Protocols
Description: Scale developed for study to quantitatively assess the number of facilitators and barriers to recruitment and testing
Time Frame: Sustainment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline assessment period, up to 2 weeks
Arm/Group | Chain Referral | Credible Messenger
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/223
Serious Adverse Events (participants affected / at risk) | 0/263 | 0/223
Other Adverse Events (participants affected / at risk) | 32/263 | 25/223
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chain Referral (N=263) | Credible Messenger (N=223)
suicidal ideation (Psychiatric disorders) | 32 (32) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT04873401/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04873401/ICF_001.pdf